CLINICAL TRIAL: NCT05925010
Title: Does Soluble Fiber Supplementation Result in Lower Postprandial Blood Glucose in Women With Gestational Diabetes Compared With no Supplementation After a Standardized Breakfast? A Randomized, Controlled, Open-label, Prospective, Monocentric Clinical Cross-over Pilot Study at the Landesklinikum Mödling.
Brief Title: Does Soluble Fiber Supplementation Result in Lower Postprandial Blood Glucose in Women With Gestational Diabetes Compared With no Supplementation After a Standardized Breakfast?
Acronym: DiFiGDM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Collaborators: Mödling Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GS1-EK-4/809-2022
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-02

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes; soluble fibre; dietary fibre; guar
MeSH Terms: conditions — Diabetes, Gestational | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplementation with soluble fibre from guar (Experimental): In the intervention group, the patients consume the standardized meal instead of breakfast and add 10 g of soluble fiber in the form of Optifibre (food for special medical purposes) to this cereal porridge.
  Interventions: Dietary Supplement: Supplementation with soluble fibre from guar (Optifibre©)
- No supplementation with soluble fibre from guar (No Intervention): In the control group, the patients eat the standardized meal without adding soluble fiber in the form of Optifibre.

INTERVENTIONS:
Dietary Supplement: Supplementation with soluble fibre from guar (Optifibre©) — 10g of soluble fibre from guar in the form of Optifibre© (dietary food for special medical purposes) is added to the standardized meal (Resource cereal porridge©).
  Arms: Supplementation with soluble fibre from guar

SUMMARY:
The objective of this study is to investigate the effect of supplementation of 10g soluble fiber from guar on postprandial blood glucose levels in women with gestational diabetes after consumption of a standardized meal compared with no supplementation.

Null Hypothesis H0:

Soluble fiber supplementation will not result in a lower postprandial blood glucose increase in women with gestational diabetes compared to no supplementation after consumption of a standardized meal.

Alternative hypothesis H1:

Soluble fiber supplementation will result in a lower postprandial blood glucose increase in women with gestational diabetes compared to no supplementation after consumption of a standardized meal.

Study participants are randomly assigned to the intervention (consumption of a standardized meal and 10g soluble fibre) or control group (consumption of a standardized meal without soluble fibre). After a 2-day wash-out phase, the two groups are switched (the intervention group becomes the control group and vice versa) with the same standardized procedure.

DETAILED DESCRIPTION:
Background and study aims:

The effect of supplementation of soluble dietary fiber from guar in the form of a dietary food for special medical purposes (Optifibre©) on postprandial glucose levels in women with gestational diabetes after a standardized test meal (Resource cereal porridge©) was consumed with or without supplementation is being investigated.

The aim of this study is to verify whether the use of easily tolerated soluble dietary fiber in addition to nutritional therapy for gestational diabetes can lead to an improvement in glycemic control and thus represent a therapeutic option for diabetic diseases in the future.

Participants:

Women with gestational diabetes meeting the inclusion criteria.

Study drain:

Study participants are recruited via the appointment at the metabolic outpatient clinic of the Mödling district, where diabetes and nutrition training including training on the Contour Next One© blood glucose meter takes place as standard.

If patients meet the inclusion criteria for participation in the study, the nutritional training is followed by an educational interview including signing of the consent form if the patient wishes to participate. After a one-week run-in phase, the participating patients are assigned to the intervention or control group by means of a randomizer. After a 2-day wash-out phase, the two groups are switched (the intervention group becomes the control group and vice versa) with the same standardized procedure.

The procedure is as follows: at the initial appointment in the metabolic outpatient clinic, the participant receives 2 sachets of a standardized cereal porridge, which represents the standardized breakfast, and 1 can of Optifibre©.

In the control phase, the participant consumes the cereal porridge with 200ml of milk after fasting blood glucose is measured. 1 hour after consumption, the postprandial blood glucose value is measured and documented in self-monitoring.

In the intervention phase, participants also replace breakfast with the same porridge, but consume an additional 10g of Optifibre© mixed into the porridge. As in the control phase, fasting blood glucose is measured beforehand and postprandial blood glucose is measured 1 hour after consumption, including documentation.

Intervention and control phase take place consecutively after a wash-out phase of 2 days. During the wash-out phase, the general guidelines for nutrition in gestational diabetes will be followed, no supplementation with Optifibre© will be given.

Participants send the records to difi.gdm@moedling.lknoe.at , the data are then pseudonymized and further processed with the appropriate verification code.

The intervention itself lasts approximately 2 weeks per participant starting with initial training and ending with the transmission of the data.

The total duration of the study is significantly longer, as recruitment is an ongoing process. It is assumed that the total duration of data collection will be at least 6 months, based on the estimate that 3 to 4 patients/week can be included and recruited for the study.

Benefits and risks:

If supplementation of the soluble fiber Guar shows a positive effect on glycemic control of a GDM, consumption of supplements such as Optifibre© represents another option for additional fiber intake and another therapeutic option for diabetic diseases in the future.

There is no disadvantage for the participants in this study. All study participants receive the same nutritional medical training that is also given to non-study participants, and there is no different treatment of the subjects during the course of the study, since each subject undergoes both the intervention and control phases.

Place where the study will be conducted:

This study is conducted by the Landesklinikum Mödling in cooperation with the Medical University of Graz.

Duration and schedule:

The concept submission took place in May 2022 and the study will be completed in July 2023.

Funding of the study:

As this is a final thesis of the university course "Applied Nutritional Medicine" at the Medical University of Graz to obtain the Master of Science of applied nutritional medicine, there is no funding involved.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with GDM by a pathological OGTT.
* Second (13th to 28th week of pregnancy) and/or third trimester (29th to 40th week of pregnancy).
* Sufficient knowledge of German to perform self-monitoring correctly
* No intolerance to standardised meals (cereal porridge) or BST supplements
* No concomitant disease requiring special dietary management

Exclusion Criteria:

* Existing diabetes mellitus type 1 or type 2 in pregnancy
* First trimester of pregnancy
* Intolerance/contraindications to any of the ingredients of Resource cereal© or Optifibre©.
* Insufficient language skills to perform self-monitoring
* Insufficient language skills to adequately implement study procedure/intervention

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The subject of the study is gestational diabetes, which is why only women are included in the study.
Enrollment: 67 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
postprandial blood glucose | 4 days
  postprandial blood glucose value in mg/dl with and without intervention

SECONDARY OUTCOMES:
difference between fasting blood glucose value and postprandial blood glucose value | 4 days
  difference between fasting blood glucose value and postprandial blood glucose value in mg/dl with and without intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Landesklinikum Mödling, Mödling, Lower Austria, Austria